CLINICAL TRIAL: NCT03551236
Title: Variability of Impedance Pneumography Tidal Breathing Flow-volume Curves During Sleep in Healthy Children
Status: Completed | Type: Observational
Sponsor: Revenio Research (Industry)
Collaborators: Children's Hospital Srebrnjak (Other)
Responsible Party: Sponsor
Other Study IDs: VCS-001
Record Dates: First submitted 2018-05-28; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study for the assessment of normal overnight variation in small healthy children using the Ventica Lung Function Testing System. The study is carried out to establish reference ranges for overnight lung function variation using the Ventica test, and to assess the impact of the demographic factors on the Ventica results.

ELIGIBILITY:
Inclusion Criteria:

* 18 months-6 years, both sexes
* Healthy at the time of inclusion
* Laboratory analyses in the reference range or not clinically relevant according to the investigator judgement
* Lung function in the reference range with a negative bronchodilator test result
* Signed informed consent

Exclusion Criteria:

* Preterm birth
* Chronic respiratory disorder of prematurity
* Recurrent bronchitis or recurrent hospitalizations because of a respiratory illness (recurrent pneumonia)
* Primary immunodeficiency
* Chronic rhinosinusitis, synonasal polyposis
* Nasal congestion, adenotonsillar hypertrophy, signs and symptoms of sleep apnea or sleep disordered breathing
* Acute respiratory infection or hospitalization because of an acute illness within 4 weeks prior to inclusion
* Personal or family history or clinical evidence of asthma, atopy or other chronic respiratory disorders (high risk for asthma and allergy)
* Use of asthma rescue or maintenance medication within 4 weeks prior to inclusion
* Implanted or external active medical devices such as pacemakers

Age Groups: Child, Adult, Older Adult
Study Population: Young children screened to have small probability of asthma or wheezing
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Normal range of variables of tidal breathing flow-volume curves (CSRmin, NLmin, etc.) | 1-3 nights per subject
  Analyse the normal range of variables that describe the shape and variability of tidal breathing flow-volume curves during natural night sleep obtained with impedance pneumography

CONTACTS AND LOCATIONS:
Overall Officials: Davor Plavec, MD, PhD, Principal Investigator — Children's Hospital Srebrnjak
Locations (1):
- Children's Hospital Srebrnjak, Zagreb, Croatia